CLINICAL TRIAL: NCT06274619
Title: Novel Mucosal Correlates Of RSV Protection In Older Adults (A Controlled Human Infection Study With RSV in Older People)
Brief Title: Novel Mucosal Correlates Of RSV Protection In Older Adults
Acronym: CHIRP01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23HH8541; MISP 59717 (Other Grant/Funding Number: MSD); 57276 (Registry Identifier: CPMS); 324970 (Other: IRAS)
Record Dates: First submitted 2024-02-16; First posted 2024-02-23 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteers (Experimental): Healthy volunteers aged 65-75 years undergoing controlled human infection with RSV Memphis 37
  Interventions: Biological: RSV A Memphis 37

INTERVENTIONS:
Biological: RSV A Memphis 37 — RSV A Memphis 37 challenge agent

SUMMARY:
Respiratory syncytial virus (RSV) is one of the most common causes of chest infection worldwide. Despite this, it remains an underappreciated health problem, with the first effective RSV vaccines only approved by the FDA in May 2023 and unlikely to be widely available for some time. Although RSV infection is most frequent in young children, most deaths occur in older adults, particularly in those with underlying heart and lung disease. This is believed to be due in part to the ageing immune system's reduced ability to protect against infection and symptomatic disease.

However, little is known about the way human immune responses to RSV infection in older individuals differ from those of younger people. Further understanding of the mechanisms underlying immunity and potential impairments in these higher-risk people are therefore necessary. This project aims to study the factors that influence whether or not older people develop symptomatic RSV disease in healthy older volunteers after being given an RSV-induced common cold. Samples will be taken from the blood and nose in order to identify changes in the immune system associated with susceptibility or protection in older adults. Participants will be carefully screened to ensure there are no underlying health problems that might make them more at risk of severe disease and will be monitored closely throughout the course of infection. It is anticipated that differences in immune markers in the nose and/or blood of healthy older people will predict whether or not such individuals become infected or develop symptoms. By analysing the networks of genes that are switched on and off, the aim is to identify the pathways in the immune system responsible for these differences, to ultimately develop improved diagnostic tests, vaccines and treatments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons aged 65 to 75 years, able to give informed consent
* Non-smokers or ex-smokers with a pack year history of 10 or less
* Spirometry within the normal range for age and height (+/- 15%)
* Forced Expiratory Volume / Forced Vital Capacity (FEV1/FVC) >70% without bronchodilator
* Vaccination against severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at the minimum of 4 weeks prior to screening

Exclusion Criteria:

* Chronic respiratory disease (asthma, chronic obstructive pulmonary disease, rhinitis, sinusitis) in adulthood
* Inhaled bronchodilator or steroid use within the last 12 months
* Habitual use of any medication or other product (prescription or over the counter) for symptoms of rhinitis or nasal congestion within the last 3 months
* Acute upper respiratory infection (URI or sinusitis) in the past 6 weeks
* Participants with allergic symptoms present at baseline
* Clinically relevant abnormality on chest X-ray
* Those in close domestic contact (i.e. sharing a household with, caring for, or daily face to face contact) with children under 3 years, clinically vulnerable and/or immunosuppressed persons, or those with chronic respiratory disease
* Participants with known or suspected immune deficiency
* Receipt of systemic glucocorticoids (in a dose ≥ 5 mg prednisone daily or equivalent) within one month, or any other cytotoxic or immunosuppressive drug within 6 months prior to challenge
* Known Immunoglobulin A (IgA) deficiency, immotile cilia syndrome, or Kartagener's syndrome
* History of frequent nose bleeds
* Any significant medical condition or prescribed drug deemed by a study doctor to make the participant unsuitable for the study
* Recent or current use of recreational drugs, confirmed by a positive urine drug screen
* History of difficult blood draw, syncope or poor tolerance of sampling procedures

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of solicited and unsolicited adverse events (AEs) | 28 Days
  Number of solicited and unsolicited adverse events (AEs) from virus inoculation (Day 0) to Day 28 post-inoculation
Infection rate | 10 days
  Infection rate calculated by the number of infected individuals over the number of uninfected individuals expressed as a percentage, with infection defined as 2 or more quantifiable greater than lower limit of quantification (viral load ≥LLOQ) by RT-PCR from nasal wash, reported on 2 or more consecutive timepoints, starting from Day 2 post-inoculation and up to discharge from quarantine

SECONDARY OUTCOMES:
Nasal Viral Load | 28 days
  Mean nasal viral load by reverse transcription polymerase chain reaction (RT-PCR) reported in Log10 copies/mL
Antibody levels by serum neutralisation assay | 28 days
  Antibody levels in blood by serum neutralisation assay by Log2 Geometric Mean Titre
Antibody levels by ELISA | 28 days
  Antibody levels in blood by Enzyme-linked immunosorbent assay (ELISA) by Log2 Geometric Mean Titre

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Chiu, Principal Investigator — Imperial College London
Locations (1):
- Imperial Clinical Research Facility, Imperial College Healthcare NHS Trust, London, United Kingdom